CLINICAL TRIAL: NCT04125641
Title: Non-Interventional Study on Effectiveness of Elxaban Tab. in Patients With Non-valvular Atrial Fibrillation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2019-0536
Record Dates: First submitted 2019-10-07; First posted 2019-10-14 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Atrial Fibrillation
Keywords: Elxaban
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elxaban group: AF patients taking Elxaban

SUMMARY:
This study is prospective Cohort study which was performed in multicenter (General Hospital) in Korea. Inclusion criteria is patients with atrial fibrillation taking Elxaban (generic drug of apixaban) who visit hospital. The purpose is to analyze bleeding (major bleeding, minor bleeding), stroke, systemic embolism, death, other clinical events (acute myocardial infarction, pulmonary embolism, transient ischemic attack, hospitalization), drug adherence, questionnaire of life quality (AFEQT), cognitive function (KDSQ) according to the use of Elxaban.

ELIGIBILITY:
Inclusion Criteria:

1. patients with atrial fibrillation taking Elxaban (patients with age more than 19)
2. Patients who agree with study inclusion

Exclusion Criteria:

1. patients who do not agree with study inclusion
2. patients with age less than 19
3. Pregnancy, Breastfeeding

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Atrial fibrillatin patients taking Elxaban in general hospital
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-01-02 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
major bleeding | 1 month
  Major bleeding is defined according to the criteria of the International Society on Thrombosis and Haemostasis (ISTH).
  1. Fatal bleeding, and/or
  2. Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarticular or pericardial, or intramuscular with compartment syndrome, and/or
  3. Bleeding causing a fall in hemoglobin level of 20 g/L (1.24 mmol/L) or more, or leading to transfusion of two or more units of whole blood or red cells.
major bleeding | 6 months
  Major bleeding is defined according to the criteria of the International Society on Thrombosis and Haemostasis (ISTH).
  1. Fatal bleeding, and/or
  2. Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarticular or pericardial, or intramuscular with compartment syndrome, and/or
  3. Bleeding causing a fall in hemoglobin level of 20 g/L (1.24 mmol/L) or more, or leading to transfusion of two or more units of whole blood or red cells.
major bleeding | 12 months
  Major bleeding is defined according to the criteria of the International Society on Thrombosis and Haemostasis (ISTH).
  1. Fatal bleeding, and/or
  2. Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarticular or pericardial, or intramuscular with compartment syndrome, and/or
  3. Bleeding causing a fall in hemoglobin level of 20 g/L (1.24 mmol/L) or more, or leading to transfusion of two or more units of whole blood or red cells.
major bleeding | 24 months
  Major bleeding is defined according to the criteria of the International Society on Thrombosis and Haemostasis (ISTH).
  1. Fatal bleeding, and/or
  2. Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarticular or pericardial, or intramuscular with compartment syndrome, and/or
  3. Bleeding causing a fall in hemoglobin level of 20 g/L (1.24 mmol/L) or more, or leading to transfusion of two or more units of whole blood or red cells.
Stroke | 1 month
  Stroke included both ischemic and hemorrhagic stroke.
Stroke | 6 months
  Stroke included both ischemic and hemorrhagic stroke.
Stroke | 12 months
  Stroke included both ischemic and hemorrhagic stroke.
Stroke | 24 months
  Stroke included both ischemic and hemorrhagic stroke.
systemic embolism | 1 month
  An SEE(systemic embolism) was defined by both clinical and objective evidence of sudden loss of end-organ perfusion
systemic embolism | 6 months
  An SEE(systemic embolism) was defined by both clinical and objective evidence of sudden loss of end-organ perfusion
systemic embolism | 12 months
  An SEE(systemic embolism) was defined by both clinical and objective evidence of sudden loss of end-organ perfusion
systemic embolism | 24 months
  An SEE(systemic embolism) was defined by both clinical and objective evidence of sudden loss of end-organ perfusion
death | 1 month
  Death included overall death, cardiovascular death and non-cardiovascular death.
death | 6 months
  Death included overall death, cardiovascular death and non-cardiovascular death.
death | 12 months
  Death included overall death, cardiovascular death and non-cardiovascular death.
death | 24 months
  Death included overall death, cardiovascular death and non-cardiovascular death.

SECONDARY OUTCOMES:
other clinical events: acute myocardial infarction | 1 month
  Myocardial infarction (MI) is defined as a clinical (or pathologic) event in the setting of myocardial ischemia in which there is evidence of myocardial injury. The diagnosis is secured when there is a rise and/or fall of troponin (high sensitivity assays are preferred) along with supportive evidence in the form of typical symptoms, suggestive electrocardiographic (ECG) changes, or imaging evidence of new loss of viable myocardium or new regional wall motion abnormality.
other clinical events: acute myocardial infarction | 6 months
  Myocardial infarction (MI) is defined as a clinical (or pathologic) event in the setting of myocardial ischemia in which there is evidence of myocardial injury. The diagnosis is secured when there is a rise and/or fall of troponin (high sensitivity assays are preferred) along with supportive evidence in the form of typical symptoms, suggestive electrocardiographic (ECG) changes, or imaging evidence of new loss of viable myocardium or new regional wall motion abnormality.
other clinical events: acute myocardial infarction | 12 months
  Myocardial infarction (MI) is defined as a clinical (or pathologic) event in the setting of myocardial ischemia in which there is evidence of myocardial injury. The diagnosis is secured when there is a rise and/or fall of troponin (high sensitivity assays are preferred) along with supportive evidence in the form of typical symptoms, suggestive electrocardiographic (ECG) changes, or imaging evidence of new loss of viable myocardium or new regional wall motion abnormality.
other clinical events: acute myocardial infarction | 24 months
  Myocardial infarction (MI) is defined as a clinical (or pathologic) event in the setting of myocardial ischemia in which there is evidence of myocardial injury. The diagnosis is secured when there is a rise and/or fall of troponin (high sensitivity assays are preferred) along with supportive evidence in the form of typical symptoms, suggestive electrocardiographic (ECG) changes, or imaging evidence of new loss of viable myocardium or new regional wall motion abnormality.
other clinical events: pulmonary embolism | 1 month
  Pulmonary embolism is defined as sudden closure of a pulmonary artery or one of its branches, caused by a blood-borne clot or foreign material that plugs the vessel.
other clinical events: pulmonary embolism | 6 months
  Pulmonary embolism is defined as sudden closure of a pulmonary artery or one of its branches, caused by a blood-borne clot or foreign material that plugs the vessel.
other clinical events: pulmonary embolism | 12 months
  Pulmonary embolism is defined as sudden closure of a pulmonary artery or one of its branches, caused by a blood-borne clot or foreign material that plugs the vessel.
other clinical events: pulmonary embolism | 24 months
  Pulmonary embolism is defined as sudden closure of a pulmonary artery or one of its branches, caused by a blood-borne clot or foreign material that plugs the vessel.
other clinical events: transient ischemic attack | 1 month
  Transient ischemic attack (TIA, Mini-Stroke) is defined as a neurological event with the signs and symptoms of a stroke, but which go away within a short period of time.
other clinical events: transient ischemic attack | 6 months
  Transient ischemic attack (TIA, Mini-Stroke) is defined as a neurological event with the signs and symptoms of a stroke, but which go away within a short period of time.
other clinical events: transient ischemic attack | 12 months
  Transient ischemic attack (TIA, Mini-Stroke) is defined as a neurological event with the signs and symptoms of a stroke, but which go away within a short period of time.
other clinical events: transient ischemic attack | 24 months
  Transient ischemic attack (TIA, Mini-Stroke) is defined as a neurological event with the signs and symptoms of a stroke, but which go away within a short period of time.
drug adherence | 1 month
  Drug adherence is defined as the extent to which a patient takes his or her medication as prescribed
drug adherence | 6 months
  Drug adherence is defined as the extent to which a patient takes his or her medication as prescribed
drug adherence | 12 months
  Drug adherence is defined as the extent to which a patient takes his or her medication as prescribed
drug adherence | 24 months
  Drug adherence is defined as the extent to which a patient takes his or her medication as prescribed
questionnaire of life quality (AFEQT) | 1 month
  AFEQT is a validated questionnaire that was patient derived with expert clinical input, and is easy to use format with 20 questions on a seven point Likert scale. AFEQT evaluates Health Related Quality of Life (HRQoL) across three domains
  * Symptoms - Four questions specifically targeted to assess AF related symptoms
  * Daily Activities - Eight questions that evaluate daily function in AF patients
  * Treatment Concerns - Six questions that assess AF treatment concerns in patients
    * Scoring key provides information on how to score the questionnaire and explains how to interpret results. The scoring key provides the following scores:•Overall AFEQT Score (18 questions) •Treatment Satisfaction Score (2 questions)
questionnaire of life quality (AFEQT) | 6 months
  AFEQT is a validated questionnaire that was patient derived with expert clinical input, and is easy to use format with 20 questions on a seven point Likert scale. AFEQT evaluates Health Related Quality of Life (HRQoL) across three domains
  * Symptoms - Four questions specifically targeted to assess AF related symptoms
  * Daily Activities - Eight questions that evaluate daily function in AF patients
  * Treatment Concerns - Six questions that assess AF treatment concerns in patients
    * Scoring key provides information on how to score the questionnaire and explains how to interpret results. The scoring key provides the following scores:•Overall AFEQT Score (18 questions) •Treatment Satisfaction Score (2 questions)
questionnaire of life quality (AFEQT) | 12 months
  AFEQT is a validated questionnaire that was patient derived with expert clinical input, and is easy to use format with 20 questions on a seven point Likert scale. AFEQT evaluates Health Related Quality of Life (HRQoL) across three domains
  * Symptoms - Four questions specifically targeted to assess AF related symptoms
  * Daily Activities - Eight questions that evaluate daily function in AF patients
  * Treatment Concerns - Six questions that assess AF treatment concerns in patients
    * Scoring key provides information on how to score the questionnaire and explains how to interpret results. The scoring key provides the following scores:•Overall AFEQT Score (18 questions) •Treatment Satisfaction Score (2 questions)
questionnaire of life quality (AFEQT) | 24 months
  AFEQT is a validated questionnaire that was patient derived with expert clinical input, and is easy to use format with 20 questions on a seven point Likert scale. AFEQT evaluates Health Related Quality of Life (HRQoL) across three domains
  * Symptoms - Four questions specifically targeted to assess AF related symptoms
  * Daily Activities - Eight questions that evaluate daily function in AF patients
  * Treatment Concerns - Six questions that assess AF treatment concerns in patients
    * Scoring key provides information on how to score the questionnaire and explains how to interpret results. The scoring key provides the following scores:•Overall AFEQT Score (18 questions) •Treatment Satisfaction Score (2 questions)
cognitive function (KDSQ) | 1 month
  The KDSQ consists of three subscales (i.e., global memory function, other cognitive function, and instrumental activities of daily living), including 15 items that can detect early changes in cognitive decline to diagnose dementia.
cognitive function (KDSQ) | 6 months
  The KDSQ consists of three subscales (i.e., global memory function, other cognitive function, and instrumental activities of daily living), including 15 items that can detect early changes in cognitive decline to diagnose dementia.
cognitive function (KDSQ) | 12 months
  The KDSQ consists of three subscales (i.e., global memory function, other cognitive function, and instrumental activities of daily living), including 15 items that can detect early changes in cognitive decline to diagnose dementia.
cognitive function (KDSQ) | 24 months
  The KDSQ consists of three subscales (i.e., global memory function, other cognitive function, and instrumental activities of daily living), including 15 items that can detect early changes in cognitive decline to diagnose dementia.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology Severance Cardiovascular Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No